CLINICAL TRIAL: NCT04656704
Title: Investigating Hyaluronidase in Treating Oral Microstomia in Patients With Sclerosing Skin Disease
Brief Title: Hyaluronidase in Treating Oral Microstomia in Patients With Sclerosing Skin Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI no longer pursuing clinical trial
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Avery LaChance, Attending Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003096
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Microstomia; Scleroderma; CREST Syndrome; Scleromyxedema; Morphea
MeSH Terms: conditions — Microstomia; Scleroderma, Diffuse; CREST Syndrome; Scleromyxedema; Scleroderma, Localized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyaluronidase 200mg monthly (Experimental): Hyaluronidase 200mg monthly (Weeks 0, 4, 8, 12, 16, 20); for six doses; a 6-month treatment course with follow-up 1 month after
  Interventions: Drug: hyaluronidase injected intradermally

INTERVENTIONS:
Drug: hyaluronidase injected intradermally — Patients will receive 200 units of hyaluronidase injected intradermally to the cutaneous lips on Weeks 0, 4, 8, 12, and 16, and 20

SUMMARY:
The principal objective is to measure the degree to which oral microstomia caused by sclerosing skin disease improves after treating patients with local hyaluronidase injections. Investigator will determine improvements in oral aperture by measuring the centimeters of the height of oral opening.

The secondary objectives are: Investigator will aim to assess changes in quality of life and functionality, by serial calculations of the Mouth Handicap in Systemic Sclerosis (MHISS). In addition, investigator would like to investigate how many treatments are required prior to treatment efficacy plateauing. Since there is minimal data on the use of hyaluronidase for oral microstomia, it is not yet clear how many treatments are ideally required for maximal effect.

Patients will be brought in monthly for photographs, examination, assessment, and treatment.

Our hypothesis is that hyaluronidase injections will significantly improve patients' ability to open their mouths and oral functionality. It remains unclear how many treatments will be required for maximal effect.

DETAILED DESCRIPTION:
Investigator will recruit 8 patients with oral microstomia caused by a sclerotic skin disorder. Patients must be 18 years of age or older with an established diagnosis of a sclerotic skin disorder by a dermatologist. Sclerotic skin disorders may include scleroderma, CREST, scleromyxedema, and morphea involving the face.

At the initial screening visit, demographic information will be obtained, inclusion and exclusion criteria will be reviewed, and informed consent will be obtained for those deemed eligible for enrollment. Patients who qualify for the study, and who have never been exposed to hyaluronidase before, will have 0.1 cc hyaluronidase injected to assess whether they have an allergic reaction.

Qualifying patients will undergo monthly intradermal injections of 200 units of hyaluronidase into the cutaneous lips by the study staff into through 6 treatments. Subjects will be evaluated for improvement in primary and secondary endpoints using clinical examination, photographs, and questionnaires during initial and follow-up visits.

Since this is a pilot study, there are only 2 case reports published wherein hyaluronidase was used for similar indications. One study injected approximately between 120 and 150 units for morphea-induced microstomia; this study listed locations of injection sites (ie, right jaw line, left jawline, and chin). Another used between 20 and 200 units of hyaluronidase for scleroderma-induced microstomia; investigators injected in 2 rows of the cutaneous lips and approximated number of injections in a schematic. Investigator elected to inject the higher end of dosage used, 200 units (1 full vial of hyaluronidase), as this was effectively used in a publication. Additionally, there has not been any dose-related side effect concerns with hyaluronidase to our knowledge. It is common practice to use multiple vials to treat hyaluronic acid complications, which is safely done.

Subjects will be evaluated for improvement in primary and secondary endpoints using clinical examination, photographs, and questionnaires during initial and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Established diagnosis of a sclerosing skin disease (i.e., systemic sclerosis, CREST, scleromyxedema, morphea) by a dermatologist
3. Ability and willingness to provide informed consent, participate in study visits, and undergo visit procedures
4. Symptoms are not resolved by current treatment

Exclusion Criteria:

1. Prior treatment with hyaluronidase for oral microstomia
2. Treatment with hyaluronic acid soft tissue filler in perioral region within the last 1.5 years
3. Treatment with any semi-permanent or permanent soft tissue filler in the perioral region in the last 3 years
4. New treatment initiation (within 3 months) with immune-regulating medication, including methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, intravenous immunoglobulins, systemic steroids, or rituximab
5. New initiation of physical/occupational therapy for muscles of the face within the last 3 months
6. Known hypersensitivity to hyaluronidase
7. Women of reproductive potential who are or plan to become pregnant or breastfeed during study participation or are unable or not willing to use birth control during the study. Options for birth control include abstinence, double barrier (i.e. male condom and female diaphragm), vasectomy, intrauterine device, and hormonal contraception. Females who have not had menses within 1 year of the baseline, bilateral tubal ligation, hysterectomy, and/or bilateral oophorectomy do not require additional methods of contraception during study participation
8. Unstable condition or status, as per study investigator's judgment, that may lead to more likely discontinuation from the study including, but are not limited to, major, recurrent medical illnesses that may require hospital admission, and/or inability to participate in all study visits
9. Concurrent topical steroid use during the study (Note: topical steroid use up until the start of the study enrollment is allowed and no washout period will be required)
10. Concurrent ingestion of high dose salicylates, cortisone, ACTH, estrogens, or antihistamines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of oral aperture at the largest diameter | Weeks 0, 4, 8, 12, 16, 20, and 24
  Change of oral aperture at the largest diameter, in centimeters, with the patient's mouth opened as widely as possible. Measurements will be completed by study personnel.